CLINICAL TRIAL: NCT00590252
Title: Clinical Testing of New MR Pulse Sequences
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Frank John Rybicki, MD, PhD, Director, Cardiac CT and Vascular CT and MRI, Brigham and Women's Hospital
Other Study IDs: 2001-P-000545
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: The Focus of This Study Are New Pulse Sequences.
Keywords: Magnetic Resonance; Imaging; Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — There are no biospecimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Scheduled for an MRI: Clinically Indicated Adults

SUMMARY:
To test and validate newly developed magnetic resonance (MR) pulse sequences for their ability to enhance the collection of morphological, biomedical, and functional information from the human body. To test clinical protocols on the various MR systems available at Brigham and Women's Hospital (BWH).

DETAILED DESCRIPTION:
Magnetic resonance (MR) scanners use computer software, called pulse sequences, to extract different types of information from the human body. Though MR has largely matured to become a routine clinical imaging modality, substantial development is still underway in order to fully exploit the technology. BWH Radiology has been a leader in pulse sequence development and the protocol under review has played a large part in this development over the last several years.

The importance of further development in MR cannot be understated. In particular, biochemical information, detailed properties of water diffusion and perfusion in tissue, cardiac imaging, and high-resolution brain imaging, all hold great potential for improving medical diagnosis and monitoring.

MR pulse sequence software is typically developed in small incremental steps. For example, an investigator may receive a new state of the art sequence from the manufacturer of the scanner equipment. (S)he may then decide to add flow-sensitizing gradients. This process is not straightforward, but requires extensive testing, first in phantoms and then in-vivo, to determine if the pulse sequence is capable of performing the new task and, moreover, to see if the new feature does not introduce undesired artifacts.

Some modifications, like the introduction diffusion-sensitizing gradients, must be tested in patients, since changes of tissue diffusion can only be observed in stroke victims. Once the researcher attained the first goal, (s)he may proceed with other modifications, e.g., modifications which will improve the temporal resolution. The completion of a new sequence, which ultimately may be used in a large normal subject or patient study, may involve a large number of design steps, where each step must be tested in one or a few subjects before development proceeds. Another scenario is the application of an existing patient protocol to different, existing, and FDA approved equipment. For example the need may arise to use a different radiofrequency coil (surface coil instead of head coil) or a scanner system with different magnetic field strength (3.0 Tesla instead of 1.5 Tesla). Several parameters, such as signal-to-noise ratio, or T1 and T2 weighting may change under such circumstances. In most cases only a study in a subject will reveal if protocol parameter settings are adequate. Therefore, this protocol is different from a conventional study, where exactly the same protocol will be applied to each of a large number of subjects. However, the protocol and the general procedures of data handling used during the different scans is similar enough, so it can be summarized into a general development protocol.

The purpose of this protocol is to test and validate newly developed MR pulse sequences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Patients undergoing clinical indicated MRI

Exclusion Criteria:

* Patients with contraindication for MRI
* Pregnant women will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Rybicki, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Mulkern RV, Barnes AS, Haker SJ, Hung YP, Rybicki FJ, Maier SE, Tempany CM. Biexponential characterization of prostate tissue water diffusion decay curves over an extended b-factor range. Magn Reson Imaging. 2006 Jun;24(5):563-8. doi: 10.1016/j.mri.2005.12.008. Epub 2006 Feb 20. PMID 16735177
- [Background] Ersoy H, Goldhaber SZ, Cai T, Luu T, Rosebrook J, Mulkern R, Rybicki F. Time-resolved MR angiography: a primary screening examination of patients with suspected pulmonary embolism and contraindications to administration of iodinated contrast material. AJR Am J Roentgenol. 2007 May;188(5):1246-54. doi: 10.2214/AJR.06.0901. PMID 17449767
- [Background] McDannold N, Barnes AS, Rybicki FJ, Oshio K, Chen NK, Hynynen K, Mulkern RV. Temperature mapping considerations in the breast with line scan echo planar spectroscopic imaging. Magn Reson Med. 2007 Dec;58(6):1117-23. doi: 10.1002/mrm.21322. PMID 18046702